CLINICAL TRIAL: NCT01635361
Title: Understanding and Appraising the New Medicine Service in England
Acronym: NMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Department of Health, United Kingdom (Other Government); University College, London (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12024
Record Dates: First submitted 2012-06-19; First posted 2012-07-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Hypertension; Blood Coagulation
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Hypertension; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMS (Experimental): Patients in this arm will receive the full NMS service
  Interventions: Other: New Medicine Service
- Current Practice (No Intervention): Patients in this arm will receive the normal advice with their new medicine as dictated by current professional practice

INTERVENTIONS:
Other: New Medicine Service — The New Medicine Service is an intervention where patients prescribed a new medicine receive followup consultations with the pharmacist 7-14 days and 14-21 days after receiving the new prescription item
  Arms: NMS

SUMMARY:
About 25% medicines prescribed for long term conditions are not taken as directed, and approximately 15% people receiving a new medicine take few, if any, doses. The New Medicine Service (NMS) is a community pharmacy service that started in England in October 2011 which involves the pharmacist providing additional support to patients starting a new medicine for some breathing problems (asthma & COPD), high blood pressure, adult onset diabetes or medicines which reduce blood clotting. It aims to improve the way patients take their medicines improving outcomes and reducing costs to the National Health Service (NHS).

The investigators will assess the effectiveness and cost effectiveness of the NMS using a research study where some people will receive the NMS, and some won't, so The investigators can look at the effect of the NMS on problems with their medicines, medicines taking and use of the NHS in general. Data will be collected in the East Midlands, South Yorkshire and London areas.

The investigators will recruit 500 patients from a range of different pharmacies and follow them up at six, ten and twenty six weeks after starting their new medicine to assess effects on medicines taking behaviour, patients' reported problems with medicines, referrals to their General Practitioner (GP) and use of NHS resources. The investigators will compare the data gathered from this study with that being collected routinely by all pharmacies in England to provide wider estimates of cost effectiveness.

The investigators will also explore how the NMS service is being implemented by pharmacies. A sample of patients from the main study will be followed in more detail. This will involve recording the consultations with the pharmacist and also interviewing patients about their experience of the service. The investigators will interview the patients GP to investigate their views of the service. The investigators will also try to understand why people decline the invitation for the NMS

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling patients eligible for NMS (aged from 14 years starting a new medicine for asthma/COPD, diabetes (Type 2), antiplatelet/anticoagulation or hypertension).

Exclusion Criteria:

* Patients collecting a repeat prescription for a medicine (i.e. not new) for asthma/COPD, type 2 diabetes mellitus (T2DM), antiplatelets/anticoagulants or hypertension
* Patients collecting a medicine where the only change from the previous medicine involves a dosage or formulation change only
* Participants who are unable to understand patient/participant study documents
* Participants who are unable and unwilling to provide written consent / assent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Medicines adherence | Change in adherence from 6 weeks to 10 weeks and 26 weeks
  Patients will report medicines adherence using the service specified adherence question and against standard adherence scales
Cost effectiveness | 6 months
  Patients will record all NHS resource use during the study period via a self completion diary to assess the impact on cost effectiveness up to 6 months post initiation.
Operation of the NMS | 1 year from first recruited patient
  The investigators will qualitatively describe the operation of the NMS, the complexity and nature of resulting consultations in terms of patient engagement, advice-giving and support. Additionally it will determine acceptability to stakeholders, reasons for success or lack of success, feasibility within the service delivery environment and generalisability and replicability across disease indications and community pharmacy settings

SECONDARY OUTCOMES:
Patients' understanding of their medicines | 10 weeks
  The investigators will qualitatively evaluate patients' understanding of their medicines and the extent to which they are informed and supported in their medicines-related behaviour.
Pharmacovigilance | 1 year from first recruited patient
  The investigators will qualitatively determine whether NMS encourages improved pharmacovigilance by community pharmacists and patients.
Stakeholder experience | 1 year from first recruited patient
  The investigators will qualitatively characterise patient (and/or carer) and professional experience.
Professional relationships | 1 year from first recruited patient
  The investigators will qualitatively explore inter-professional and patient-professional relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Boyd, PhD, Study Chair — University of Nottingham; Rachel A Elliott, PhD, Study Chair — University of Nottingham; Anthony J Avery, DM, Study Director — University of Nottingham; Nicholas Barber, PhD, Principal Investigator — University College, London; Rajnikant Mehta, MSc, Study Director — University of Nottingham; Justin Waring, PhD, Study Director — University of Warwick; Antony Chuter, Study Director — Patient Involvement representative
Locations (4):
- United Kingdom (4):
  - Nottinghamshire County PCT/ County Health Partnerships, Nottingham, Notts
  - Doncaster PCT, Doncaster, South Yorkshire
  - Cambden, Barnet, Islington PCTs, London
  - Nottingham City PCT/Nottingham City Care, Nottingham

REFERENCES:
- [Derived] Elliott RA, Boyd MJ, Tanajewski L, Barber N, Gkountouras G, Avery AJ, Mehta R, Davies JE, Salema NE, Craig C, Latif A, Waring J, Chuter A. 'New Medicine Service': supporting adherence in people starting a new medication for a long-term condition: 26-week follow-up of a pragmatic randomised controlled trial. BMJ Qual Saf. 2020 Apr;29(4):286-295. doi: 10.1136/bmjqs-2018-009177. Epub 2019 Nov 15. PMID 31732700
- [Derived] Elliott RA, Tanajewski L, Gkountouras G, Avery AJ, Barber N, Mehta R, Boyd MJ, Latif A, Chuter A, Waring J. Cost Effectiveness of Support for People Starting a New Medication for a Long-Term Condition Through Community Pharmacies: An Economic Evaluation of the New Medicine Service (NMS) Compared with Normal Practice. Pharmacoeconomics. 2017 Dec;35(12):1237-1255. doi: 10.1007/s40273-017-0554-9. PMID 28776320
- [Derived] Elliott RA, Boyd MJ, Salema NE, Davies J, Barber N, Mehta RL, Tanajewski L, Waring J, Latif A, Gkountouras G, Avery AJ, Chuter A, Craig C. Supporting adherence for people starting a new medication for a long-term condition through community pharmacies: a pragmatic randomised controlled trial of the New Medicine Service. BMJ Qual Saf. 2016 Oct;25(10):747-58. doi: 10.1136/bmjqs-2015-004400. Epub 2015 Dec 8. PMID 26647412
- [Derived] Boyd M, Waring J, Barber N, Mehta R, Chuter A, Avery AJ, Salema NE, Davies J, Latif A, Tanajewski L, Elliott RA. Protocol for the New Medicine Service Study: a randomized controlled trial and economic evaluation with qualitative appraisal comparing the effectiveness and cost effectiveness of the New Medicine Service in community pharmacies in England. Trials. 2013 Dec 1;14:411. doi: 10.1186/1745-6215-14-411. PMID 24289059
- See also: NMS Study homepage — http://www.NMSevaluation.org.uk